CLINICAL TRIAL: NCT04278846
Title: Efficacy of Liposomal Bupivacaine for Prolonged Postoperative Analgesia in Patient Undergoing Breast Reconstruction With Tissue Expander
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-903
Record Dates: First submitted 2016-12-28; First posted 2020-02-20 (Actual); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Pain, Postoperative; Mammaplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DepoFoam bupivacaine (Experimental): local anesthetic
  Interventions: Drug: Depofoam bupivacaine
- Bupivacaine hydrochloride (HCl) (Active Comparator): local anesthetic
  Interventions: Drug: Bupivacaine hydrochloride (HCl)

INTERVENTIONS:
Drug: Depofoam bupivacaine — The study drug Depofoam bupivacaine will be administered into the right and/or left breast of each patient 30 minutes prior to the creation of the subpectoral muscle pocket.
  Other Names: liposomal bupivacaine, Exparel
  Arms: DepoFoam bupivacaine
Drug: Bupivacaine hydrochloride (HCl) — The study drug bupivacaine HCl will be administered into the right and/or left breast of each patient 30 minutes prior to the creation of the subpectoral muscle pocket.
  Other Names: Marcaine
  Arms: Bupivacaine hydrochloride (HCl)

SUMMARY:
Patients undergoing breast reconstruction with tissue expanders will be treated with a local anesthetic during their procedure and monitor their post-operative pain level and amount of oral pain medication taken. This information will be used to determine if liposomal bupivacaine provides better and longer pain control vs. bupivacaine HCl.

DETAILED DESCRIPTION:
Fifty consecutive (25 per arm) patients undergoing unilateral or bilateral breast reconstruction with tissue expanders will be administered intraoperatively in a standardized manner with either bupivicaine HCl (control group) or liposomal bupivacaine/Exparel (experimental group). Pain will be assessed qualitatively through the use of: 1) numeric rating scale during rest (NRS-R) and activity (NRS-A), 2) brief pain inventory (BPI) questionnaire, and 3) postoperative analgesia patient satisfaction scale. Furthermore, investigators will record the use of rescue analgesics for each patient. This part of the study will provide quantitative data that investigators can then use in comparison to the qualitative measurements (NSR, BPI, patient satisfaction scale rate). In turn, this will allow us to objectify patient's pain, thereby increasing the validity of our results. More importantly, this aspect of the investigation will enable us to study the impact that liposomal bupivacaine has in reducing the postoperative usage of opioid medications in this patient population. As this is a pilot study, a sample size of 50 total patients (25 per treatment group) is planned. This sample size should provide estimates of potential effect sizes and variability in the present setting to allow for future study planning. This study should provide adequate evidence of whether pain decreases of 15% or more are unlikely in this setting.

Investigators aim to evaluate the effectiveness of DepoFoam Bupivicaine (Exparel®) to reduce postoperative pain in breast reconstruction patients compared to the current standard treatment (bupivacaine HCl). Investigators hypothesize that patients undergoing breast reconstruction with tissue expander will achieve greater control of post-operative pain and longer lasting analgesia with the use of liposomal bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* undergoing breast reconstruction with tissue expander

Exclusion Criteria:

* history of adverse reaction to local anesthesia
* chronic liver disease
* history of chronic preoperative consumption of narcotics or opioids
* history of alcohol and/or illicit drug dependence
* undergoing combined procedures
* diagnosed with neuromuscular/neurosensory disorder
* positive pregnancy test
* previous breast conservation therapy (lumpectomy with radiation treatment
* previous surgeries or trauma in the breast or chest region (denervation may bias pain perception)
* axillary node dissection
* psychosis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All eligible patients, 18 and over, undergo breast reconstruction with tissue expanders.
Enrollment: 50 (Actual)
Dates: Start 2014-08-22 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Isakov, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DepoFoam Bupivacaine; Bupivacaine HCl: local anesthetic
  Depofoam bupivacaine: The study drugs will be administered into the right and/or left breast of each patient 30 minutes prior to the creation of the subpectoral muscle pocket.
Period: Overall Study
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Started | 25 (No longer patients to study) | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The goal is to have 25 completed patients in each group. Patients that for some reason did not complete the post-operative pain assessment will be replaced.
Groups:
- Total: Total of all reporting groups
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — All eligible patients, 18 and over, undergo breast reconstruction with tissue expanders. No sex data collected, assuming all female
  Participants
    Female | 25 | 25 | 50
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The goal is to have 25 completed patients in each group. Patients that for some reason did not complete the post-operative pain assessment will be replaced.
  70 total started but dropout account for difference in overall population
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 24 | 24 | 48
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: on patients are disqualified based on data collection
  Participants
    United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: 1 Hour Pain Assessment Numeric Rating Scale During Rest
Description: Pain will be assessed qualitatively through the use of numeric rating scale (0-10) during rest (NRS-R) Scale name: Numeric rating scale during rest (NRS-R) The higher scores indicate more severe pain during rest (10 meaning the worst pain, 0 meaning no pain)
Time Frame: 1 hour post-operatively
Population: All randomized patients
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Bupivacaine HCl: local anesthetic
  bupivacaine HCl: The study drugs will be administered into the right and/or left breast of each patient 30 minutes prior to the creation of the subpectoral muscle pocket.
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 25 | 25
units on a scale | 5 [3 to 6] | 5 [3 to 6]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .87, Kruskal-Wallis

2. Primary Outcome: 8-12 Hour Pain Assessment Numeric Rating Scale During Rest
Description: Pain will be assessed qualitatively through the use of numeric rating scale (0-10) during rest (NRS-R) The higher scores indicate more severe pain during rest (10 meaning the worst pain, 0 meaning no pain)
Time Frame: 8-12 hours post-operatively
Population: All randomized patients
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Bupivacaine HCl: local anesthetic
  bupivacaine HCl: The study drug bupivacaine HCl will be administered into the right and/or left breast of each patient 30 minutes prior to the creation of the subpectoral muscle pocket.
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 25 | 25
units on a scale | 3 [2 to 4] | 3 [2 to 4]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .49, Kruskal-Wallis

3. Primary Outcome: 24 Hour Pain Assessment Numeric Rating Scale During Rest
Description: Pain will be assessed qualitatively through the use of numeric rating scale (0-10) during rest (NRS-R).
  The higher scores indicate more severe pain during rest (10 meaning the worst pain, 0 meaning no pain)
Time Frame: 24 hours post-operatively
Population: All randomized patients who completed the tools
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 23 | 24
units on a scale | 3 [2 to 5] | 3.5 [2.5 to 5]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .57, Kruskal-Wallis

4. Primary Outcome: 36 Hour Pain Assessment Numeric Rating Scale During Rest
Description: as for outcome 3
Time Frame: 36 hours post-operatively
Population: All randomized patients who completed the tools
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 25 | 24
units on a scale | 3 [2 to 5] | 3 [2 to 4]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine; Test type: Superiority; p = .3, Kruskal-Wallis

5. Primary Outcome: 48 Hour Pain Assessment Numeric Rating Scale During Rest
Description: Pain will be assessed qualitatively through the use of numeric rating scale during rest (NRS-R).
  The higher scores indicate more severe pain during rest (10 meaning the worst pain, 0 meaning no pain) The range is 0 to 10.
Time Frame: 48 hours post-operatively
Population: All patients who completed tools
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 23 | 23
units on a scale | 3 [2 to 5] | 3 [2 to 4]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .99, Kruskal-Wallis

6. Primary Outcome: 60 Hour Pain Assessment Numeric Rating Scale During Rest
Description: as for outcome 5
Time Frame: 60 hours post-operatively
Population: All patients who completed tools
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 24 | 25
units on a scale | 3 [1.5 to 4] | 2 [1 to 3]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .33, Kruskal-Wallis

7. Primary Outcome: 72 Hour Pain Assessment Numeric Rating Scale During Rest
Description: as for outcome 5
Time Frame: 72 hours post-operatively
Population: All randomized patients
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 23 | 25
units on a scale | 3 [1 to 4] | 2 [1 to 3]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .26, Kruskal-Wallis

8. Primary Outcome: 84 Hour Pain Assessment Numeric Rating Scale During Rest
Description: Pain will be assessed qualitatively through the use of numeric rating scale (0-10) during rest (NRS-R).
  The higher scores indicate more severe pain during rest (10 meaning the worst pain, 0 meaning no pain) The range is 0 to 10.
Time Frame: 84 hours post-operatively
Population: All randomized patients
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 21 | 25
units on a scale | 1 [1 to 3] | 2 [1 to 3]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .79, Kruskal-Wallis

9. Primary Outcome: 96 Hour Pain Assessment Numeric Rating Scale During Rest
Description: Pain will be assessed qualitatively through the use of numeric rating scale (0-10) during rest (NRS-R).
  The higher scores indicate more severe pain during rest (10 meaning the worst pain, 0 meaning no pain) Range 0-10
Time Frame: 96 hours post-operatively
Population: All randomized patients who completed the tools
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 20 | 24
units on a scale | 1.5 [.5 to 2] | 2 [1 to 3]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .62, Kruskal-Wallis

10. Primary Outcome: 36 Hour Pain Assessment Numeric Rating Scale During Activity
Description: Pain will be assessed qualitatively through the use of numeric rating scale (0-10) during activity (NRS-A).
  The higher scores indicate more severe pain during activity (10 meaning the worst pain, 0 meaning no pain) The range is 0 to 10.
Time Frame: 36 hours post-operatively
Population: All randomized patients who completed the tools
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 18 | 19
units on a scale | 5 [3 to 6] | 5 [3 to 7]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .94, Kruskal-Wallis

11. Primary Outcome: 48 Hour Pain Assessment Numeric Rating Scale During Activity
Description: Pain will be assessed qualitatively through the use of numeric rating scale (0-10) during activity (NRS-A).
  The higher scores indicate more severe pain during activity (10 meaning the worst pain,0 meaning no pain) The range is 0 to 10.
Time Frame: 48 hours post-operatively
Population: All randomized patients who completed the tools
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 17 | 18
units on a scale | 4 [4 to 5] | 5 [3 to 7]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .95, Kruskal-Wallis

12. Primary Outcome: 60 Hour Pain Assessment Numeric Rating Scale During Activity
Description: as for outcome 10
Time Frame: 60 hours post-operatively
Population: All randomized patients who completed the tools
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 17 | 19
units on a scale | 5 [2 to 6] | 4 [2 to 7]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .54, Kruskal-Wallis

13. Primary Outcome: 72 Hour Pain Assessment Numeric Rating Scale During Activity
Description: as for outcome 10
Time Frame: 72 hours post-operatively
Population: All randomized patients who completed the tools
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 16 | 19
units on a scale | 4 [3 to 5.5] | 4 [1 to 6]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .95, Kruskal-Wallis

14. Primary Outcome: 84 Hour Pain Assessment Numeric Rating Scale During Activity
Description: as for outcome 10
Time Frame: 84 hours post-operatively
Population: All randomized patients who completed the tools
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 15 | 19
units on a scale | 4 [2 to 5] | 3 [1 to 6]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .96, Kruskal-Wallis

15. Primary Outcome: 96 Hour Pain Assessment Numeric Rating Scale During Activity
Description: as for outcome 10
Time Frame: 96 hours post-operatively
Population: All randomized patients who completed the tools
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 14 | 18
units on a scale | 3.5 [2 to 5] | 3 [1 to 5]

16. Primary Outcome: 24 Hour Pain Assessment Brief Pain Inventory
Description: Pain will be assessed qualitatively through the use of the Brief Pain Inventory (BPI) Questionnaire This is also a validated scale from 0 to 10, with 10 having the most severe pain and 0 being no pain
Time Frame: 24 hours post-operatively
Population: All patients who used medication
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 22 | 23
units on a scale | 4 [3 to 5] | 5 [3 to 6]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .088, Kruskal-Wallis

17. Primary Outcome: 48 Hour Pain Assessment Brief Pain Inventory
Description: as for outcome 16
Time Frame: 48 hours post-operatively
Population: All participants who used medication
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 22 | 24
units on a scale | 3.5 [3 to 5] | 4 [3 to 5]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .42, Kruskal-Wallis

18. Primary Outcome: 72 Hour Pain Assessment Brief Pain Inventory
Description: as for outcome 16
Time Frame: 72 hours post-operatively
Population: All participants who used medication
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 21 | 24
units on a scale | 3 [2 to 5] | 3 [2 to 4.5]
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .88, Kruskal-Wallis

19. Primary Outcome: 96 Hour Pain Assessment Brief Pain Inventory
Description: as for outcome 16
Time Frame: 96 hours post-operatively
Population: All participants who used medication
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 22 | 25
units on a scale | 3 [2 to 4] | 2 [2 to 4]

20. Primary Outcome: 96 Hour Pain Assessment Post-Operative Analgesia Patient Satisfaction
Description: Pain will be assessed qualitatively through the use of post-operative analgesia patient satisfaction scale (0-5) The higher scores indicate more satisfied patients.( 5 would be very satisfied-less pain, 0 would indicate unsatisfied patients-more pain)
Time Frame: 96 hours post-operatively
Population: All patients using tools
Measure: Count of Participants; unit: Participants
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 20 | 22
Participants
  1 | 0 | 1
  2 | 0 | 0
  3 | 0 | 2
  4 | 9 | 11
  5 | 11 | 8
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .12, Kruskal-Wallis

21. Secondary Outcome: 24 Hour Use of Rescue Analgesic
Description: We will record the amount in milligrams and type of rescue analgesic for each patient.
Time Frame: 24 hours post operatively
Population: All patients reporting medication use
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 25 | 25
milligrams | 63.3 (29.3) | 63.9 (47.8)
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .96, t-test, 2 sided

22. Secondary Outcome: 48 Hour Use of Rescue Analgesic
Description: We will record the amount in milligrams and type of rescue analgesic for each patient.
Time Frame: 48 hours post operatively
Population: All patients reporting medication use
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 25 | 25
milligrams | 25.1 (21.5) | 23.3 (18.4)
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .76, t-test, 2 sided

23. Secondary Outcome: 72 Hour Use of Rescue Analgesic
Description: We will record the amount in milligrams and type of rescue analgesic for each patient.
Time Frame: 72 hours post operatively
Population: All patients reporting medication use
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 25 | 25
milligrams | 20.7 (22.1) | 19.9 (15.6)
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .88, t-test, 2 sided

24. Secondary Outcome: 96 Hour Use of Rescue Analgesic
Description: We will record the amount in milligrams and type of rescue analgesic for each patient.
Time Frame: 96 hours post operatively
Population: All patients reporting medication use
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 25 | 25
milligrams | 10.2 (11.4) | 7.5 (9.4)
Statistical Analysis 1: Comparison: DepoFoam Bupivacaine vs Bupivacaine HCl; Test type: Superiority; p = .37, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: The following adverse events will be evaluated: 1) nausea; 2) vomiting; 3) constipation; 4) somnolence; 5) dizziness; 6) respiratory distress. They will be assessed at 1, 4, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after the administration of the local anesthetics.
Description: No adverse events related to the study drugs
Groups:
- DepoFoam Bupivacaine; Bupivacaine HCl: local anesthetic
  Depofoam bupivacaine: The study drugs will be administered into the right and/or left breast of each patient 30 minutes prior to the creation of the subpectoral muscle pocket.
  There were no adverse events for either arm.
Arm/Group | DepoFoam Bupivacaine | Bupivacaine HCl
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT04278846/Prot_SAP_000.pdf